CLINICAL TRIAL: NCT06371352
Title: Effect of Intermittent and Continuous Theta Burst Stimulation on Sleep Quality, Sleep Propensity, Daytime Sleepiness, and Fatigue in Depression
Brief Title: Effect of Intermittent and Continuous Theta Burst Stimulation on Sleep, Daytime Sleepiness, and Fatigue in Depression
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jakub Antczak (Other)
Collaborators: Institute of Psychiatry and Neurology, Warsaw (Other)
Responsible Party: Sponsor-Investigator, Jakub Antczak, Clinical Professor, Jagiellonian University
Organization: Jagiellonian University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JagiellonianU73
Record Dates: First submitted 2024-04-08; First posted 2024-04-17 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Unipolar Depression; Bipolar Disorder
Keywords: Unipolar Depression; Bipolar Disorder; theta burst stimulation; sleep; sleepiness; fatigue; transcranial magnetic stimulation
MeSH Terms: conditions — Depressive Disorder; Bipolar Disorder; Sleepiness; Fatigue

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, sham-controlled clinical trial in parallel design
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Placebo intervention will be delivered with a sham-coil for magnetic stimulation, which looks identical and elicits similar sounds as the coil used for active stimulation, but induces only negligible magnetic field.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- iTBS over the left DLPFC (Active Comparator): Active iTBS with intensity of 120% of the resting motor threshold recorded from the right first dorsal interosseus will be administered over the left DLPFC. Therapy will include 90 sessions (three sessions in each of 20 consecutive working days - four weeks in total). In every session 900 magnetic pulses will be elicited.
  Interventions: Device: iTBS
- cTBS over the right DLPFC (Experimental): Active cTBS with intensity of 120% of the resting motor threshold recorded from the left first dorsal interosseus will be administered over the right DLPFC. Therapy will include 90 sessions (three sessions in each of 20 consecutive working days - four weeks in total). In every session 1200 magnetic pulses will be elicited.
  Interventions: Device: cTBS
- Sham stimulation (Sham Comparator): Active iTBS or cTBS will be administered over the left or right DLPFC respectively with sham coil. Therapy will include 90 sessions (three sessions in each of 20 consecutive working days - four weeks in total). In every session 900 or 1200 magnetic pulses will be elicited.
  Interventions: Device: Sham

INTERVENTIONS:
Device: iTBS — Active iTBS over the left DLPFC to induce the long term potentiation of stimulated area.
  Arms: iTBS over the left DLPFC
Device: cTBS — Active cTBS over the right DLPFC to induce the long term potentiation of stimulated area.
  Arms: cTBS over the right DLPFC
Device: Sham — Sham iTBS or cTBS over the left or right DLPFC respectively for placebo.
  Arms: Sham stimulation

SUMMARY:
Intermittent and continuous theta-burst stimulation (iTBS and cTBS respectively) are the newer modalities of transcranial magnetic stimulation with documented efficacy in treatment of depressed mood but with conflicting results regarding their efficacy in treatment of other symptoms of depression such as insomnia, daytime sleepiness and fatigue. This study will investigate the efficacy of iTBS over the left dorsolateral prefrontal cortex (DLPFC) and cTBS over the right DLPFC, compared to sham stimulation, in treatment of insomnia, daytime sleepiness and fatigue in depression.

DETAILED DESCRIPTION:
Intermittent and continuous theta-burst stimulation (iTBS and cTBS respectively) are the newer modalities of conventional repetitive transcranial magnetic stimulation (rTMS) with documented noninferiority in improving mood in depressive disorders. The effect of both modalities on other significant depression symptoms has not been studied. In this feasibility study investigators aim primarily to assess the safety and therapeutic potential of iTBS over the left dorsolateral prefrontal cortex (lDLPFC) and cTBS over the right dorsolateral prefrontal cortex (rDLPFC) on sleep quality, sleep propensity, fatigue, and daytime sleepiness in patients with major and bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* severe or moderate depressive episode (according to international classification of diseases (ICD)-10) without psychotic symptoms at the time of inclusion
* Diagnosis of major depression (F33.1 or F33.2) or bipolar disorder (F31.3 or F31.4).
* The score of the Athens Insomnia Scale five or more
* Unchanged antidepressive pharmacotherapy at least one month prior to inclusion

Exclusion Criteria:

* Contraindications to transcranial magnetic stimulation, including ferromagnetic elements in head, pregnancy and epilepsy
* Psychotic symptoms at the time of inclusion
* Suicidal ideations and/or attempts within three months prior to inclusion

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2024-05-15 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
Beck Depression Inventory 2 | Before intervention - four weeks after finishing intervention.
  Inventory consisting of 21 items measuring cognitive, affective, somatic, and vegetative symptoms of depression. Each item is scored from 0 to 3, with a higher score denoting more severe depression. Items are related to the criteria from the Diagnostic and Statistical Manual of Mental Disorders-IV. The minimum value of the total score is 0 and the maximum is 63 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Pittsburgh Sleep Quality Index | Before intervention - four weeks after finishing intervention.
  Pittsburgh Sleep Quality Index is a questionnaire to identify sleep disturbances. It consists of a combination of Likert-type and open-ended questions, which are later converted to scaled scores. Scores for each question range from 0 to 3, with higher scores indicating greater sleep disturbances. The minimum value of the total score is 0 and the maximum is 21 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.

SECONDARY OUTCOMES:
Brief Psychiatric Rating Scale | Before intervention - four weeks after finishing intervention.
  An 18-item scale assessing negative symptoms, such as emotional withdrawal (e.g. withdrawal from relations), motor slowness and blunted affect. Each item is rated from 1 to 7 with 7-point Likert scaling, where 7 means the most severe disturbance. The minimum value of the total score is 18 and the maximum is 126 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Epworth Sleepiness Scale | Before intervention - four weeks after finishing intervention.
  An eight-item scale. Each item refers to a situation such as driving a car or sitting quietly. The subject is asked to assess the chance of dosing in each situation, ranging from 0 (no chance) to 3 (dosing very likely). The minimum value of the total score is 0 and the maximum is 24 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Fatigue Assessment Scale | Before intervention - four weeks after finishing intervention.
  A 10-item scale to assess the severity of fatigue. Each item is an expression describing the fatigue, such as: "I am bored by fatigue" or "Mentally I feel exhausted". Each item is answered using a Likert-type scale ranging from 1 (never) to 5 (always). The minimum value of the total score is 10 and the maximum is 50 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Quality of Life in Depression Scale | Before intervention - four weeks after finishing intervention.
  A 34-item, self-reported scale to assess the impact of depression on the quality of life. The scale is scored binomially with higher scores indicating a lower quality of life. The minimum value of the total score is 0 and the maximum is 34 with higher scores meaning worse outcome. Change from the baseline to the measurement done after finishing intervention, to the measurement done two weeks after finishing intervention to the measurement done four weeks after finishing intervention.
Sleep propensity non-rapid eye movement 1 sleep stage | Through study completion, an average of 1 year
  A 23-channel electroencephalography (EEG), 2-channel electrooculogram (EOG) and a chin electromyogram (EMG) recorded through 45 minutes in lying position with eyes closed. The recordings will then be divided into 30 second epochs. Each epoch will be assigned to particular sleep stage or wake, according to standards of sleep staging issued by the American Academy of Sleep Medicine [Silber et al. 2007]. The difference in the latency of non-rapid eye movement 1 sleep stage (the time from light off to the first epoch of the non-rapid eye movement 1 sleep stage) before and after intervention will be assessed.
Sleep propensity non-rapid eye movement 2 sleep stage | Through study completion, an average of 1 year
  A 23-channel electroencephalography (EEG), 2-channel electrooculogram (EOG) and a chin electromyogram (EMG) recorded through 45 minutes in lying position with eyes closed. The recordings will then be divided into 30 second epochs. Each epoch will be assigned to particular sleep stage or wake, according to standards of sleep staging issued by the American Academy of Sleep Medicine [Silber et al. 2007]. The difference in the latency of non-rapid eye movement 2 sleep stage (the time from light off to the first epoch of the non-rapid eye movement 2 sleep stage) before and after intervention will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Bogdan Stefanowski, MD, Principal Investigator — Institute of Psychiatry and Neurology
Locations (1):
- Institute of Psychiatry and Neurology, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Yes
EEG, EOG, EMG recordings, scans of scales, inventories and questionnaires will be available upon request sent per e-mail to: bstefanowski@ipin.edu.pl
Supporting Information: Study Protocol, SAP
Time Frame: December 2026 - December 2030
Access Criteria: For researchers in medical sciences and medical professional upon justification of their request.

REFERENCES:
- [Background] Silber MH, Ancoli-Israel S, Bonnet MH, Chokroverty S, Grigg-Damberger MM, Hirshkowitz M, Kapen S, Keenan SA, Kryger MH, Penzel T, Pressman MR, Iber C. The visual scoring of sleep in adults. J Clin Sleep Med. 2007 Mar 15;3(2):121-31. PMID 17557422